CLINICAL TRIAL: NCT06416228
Title: Beetroot Juice Supplement for Boosting Mucosal Immunity - The NO Cold Study
Brief Title: Beetroot Juice NO Cold Study
Acronym: NCS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Southern Methodist University (Other)
Collaborators: Baylor University (Other)
Responsible Party: Principal Investigator, Thomas Ritz, Professor, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 23-108
Record Dates: First submitted 2024-04-29; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Respiratory Tract Infections; Cold Symptoms; Exhaled Nitric Oxide
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Double blinded, placebo controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participating students and assessors will be blinded to the participants' group assignment. Since students and research staff will not know whether their beetroot juice is depleted or not, treatment conditions are double-blinded (juice "shots" will be pre-labeled by study statistician with a participant number based on the pre-study randomization, so neither the staff nor the participant know the contents). Students will also be assured of full blinding of course instructors, including the PIs and Co-Is, to names of study participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Two active doses of beetroot juice (Experimental): 2 active (nitrate containing) doses of Beet-it Pro 400
  Interventions: Dietary Supplement: Beetroot juice
- One active dose of beetroot juice and one placebo dose of beetroot juice (Active Comparator): 1 active (nitrate containing) dose of Beet-it Pro 400 and one placebo (nitrate-depleted) dose of beetroot juice
  Interventions: Dietary Supplement: Beetroot juice
- Two placebo doses of beetroot juice (Placebo Comparator): 2 placebo (nitrate-depleted) doses of beetroot juice
  Interventions: Dietary Supplement: Beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — Participants will take on dose in the morning and one in the afternoon, for 7 days during their final academic examinations
  Other Names: Beet-it 400

SUMMARY:
Currently, there is a lack of evidence-based prevention strategies for respiratory infection and management of these conditions can be costly to the public. Airway nitric oxide provides a first line of defense against pathogens, and beetroot juice, a source of dietary nitrate, has been shown to elevate nitric oxide. The main objective of this project is to demonstrate that one week of supplementation with beetroot juice elevates airway nitric oxide during stressful periods in young adults and thereby can protect against respiratory viral infections.

DETAILED DESCRIPTION:
Study Title Beetroot Juice Supplement for Boosting Mucosal Immunity: The NO Cold Study

Objectives Aim 1: Demonstrate that a 7-day trial of daily beetroot juice or nitrate depleted placebo beetroot juice is feasible with acceptable retention and adherence during a period of real-life stress, using adherence monitoring of beetroot juice intake by cell phone recorded video; acceptable burdensomeness for participants and success of team coordination and study logistics should also be demonstrated.

Aim 2: Generate initial estimates of effect size for a) elevations in exhaled nitric oxide (FENO) and b) the correlation between changes in FENO and both infection reduction and cold symptom reduction (biological signature).

Aim 3: a) Examine if 2 daily doses of beetroot juice are more potent than 1 daily dose in elevating FENO, and b) investigate whether each beetroot juice dosage (1 dose and 2 doses) increases FENO more than the placebo.

Exploratory aims: Explore sex as a moderator of all the Aims. Also explore effects of competitors/inhibitors of NO (arginase, asymmetric dimethylarginine) in a) reducing FENO under stress, and b) whether beetroot juice buffers any of these potential adverse effects on FENO; c) investigate whether effects of stress cortisol, which negatively impact NO, cold symptoms, and respiratory infections, are also buffered by beetroot juice.

Design and Outcomes This is a double-blind, placebo controlled clinical trial to test the efficacy of beetroot juice as elevating airway NO, which is associated with reduced cold symptoms and respiratory viral infection rates, in undergraduate students aged 18-30.

Interventions and Duration Participants will be receiving 1 active daily dose of beetroot juice and 1 dose of nitrate-depleted placebo beetroot juice, 2 active daily doses of beetroot juice, or 2 daily doses of nitrate-depleted placebo beetroot.

Cold symptoms will be explored by questionnaire at baseline (in a low stress period during the semester) and subsequently twice during the final exam period, once at an early stage of the finals (days 1-3 of the final exam period), and once at a later stage (days 4-6). A follow-up online questionnaire packet will be administered 3 days after the last final day. FENO, sampling for viral PCR, salivary cortisol, and exhaled breath condensate will be undertaken at baseline, early finals, and late finals (in-person assessments are not feasible at follow-up, because students leave campus after finals).

Sample Size and Population The sample size is 150 students (n=66 at SMU site, n=84 at Baylor site). Female and male students 18-30 years old will be recruited from Baylor and SMU. The investigators will make an extra effort to guarantee equal representation of both genders. Participants can be from any ethnic or cultural background, as long as they can understand and read English adequately. The student population of both universities combined is diverse (28.5-38.5% minorities).

The investigators will stratify by sex and by site, to randomize participants to receiving 1 active daily dose of beetroot juice and 1 dose of nitrate-depleted placebo beetroot juice, 2 active daily doses of beetroot juice, or 2 daily doses of nitrate-depleted placebo beetroot juice (n=50 per group).

ELIGIBILITY:
Inclusion Criteria:

Individuals will be included:

* SMU or Baylor University students
* Ages of 18-30 years old.

Exclusion Criteria:

* Active smokers
* Smoking cannabis or vape
* Students with clinically significant asthma
* COPD and emphysema
* Allergic rhinitis
* High levels of exhaled nitric oxide (FENO ≥40ppb)
* Developing kidney stone
* Clinically significant heart disease
* Cerebrovascular disease
* Thyroid dysfunction
* Out-of-control diabetes
* Significant current problems with schizophrenia, psychosis, mood disorders, suicidality, and drug or alcohol dependence or abuse

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Exhaled Nitric Oxide | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  The Fraction of NO in Exhaled Breath (FENO, in ppb) will be measured with an electrochemical gas analyzer (NIOX vero).
Viral Polymerase Chain Reaction | Baseline (non-stress mid point of semester), 4-6 days into active beetroot shots (during final examination period)
  Binary positive/negative test results for a panel of viral and bacterial respiratory pathogens.
Wisconsin Upper Respiratory Symptom Survey (WURSS) | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period), 1-3 days after finishing beetroot shots (after final examinations)
  Assess symptoms of acute upper respiratory tract infections (common cold symptoms) by questionnaire
Adherence monitoring (feasibility) | Every day during active beetroot shots (Days 1-7)
  Participants will upload a cell phone video of their intake for that day to a secure cloud folder, time stamp in comparison to assigned intake windows provides measure of adherence
Burdensomeness | 1-3 days after finishing beetroot shots (after final examinations)
  Follow-up questionnaire will be administered with the online follow-up survey. It explores experience with the best mode of reminder receipt (email or text message), whether the participants guessed their condition, and how burdensome 8 aspects of the study (including daily intake, video recording, upload, questionnaires, physiological assessment) were.

SECONDARY OUTCOMES:
Acute stress | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period), 1-3 days after finishing beetroot shots (after final examinations)
  Ad-hoc acute stress rating
Cortisol | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  Cortisol, from saliva sampled with passive drool test
Perceived stress | Baseline (non-stress mid point of semester), 4-6 days into active beetroot shots (during final examination period)
  Perceived Stress Scale (PSS)
Mood | Baseline (non-stress mid point of semester), 4-6 days into active beetroot shots (during final examination period)
  Hospital Anxiety and Depression Scale (HADS)
Blood pressure (systolic and diastolic blood pressure) and heart rate | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  Measured after at least 10 min of acclimatization to the laboratory

OTHER OUTCOMES:
One-day Food Record | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  One-day food record via the Automated Self-Administered 24-Hour platform; control variable
Arginase | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  From Exhaled breath condensate or saliva, competitors/inhibitor of NO; exploratory mediator of FENO
Asymmetric dimethylarginine | Baseline (non-stress mid point of semester), 1-3 days into active beetroot shots (during final examination period), 4-6 days into active beetroot shots (during final examination period)
  From Exhaled breath condensate or saliva, competitors/inhibitor of NO; exploratory mediator of FENO

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ritz, Ph.D., Principal Investigator — Southern Methodist University; Annie Ginty, Ph.D., Study Director — Baylor University
Locations (2):
- United States (2):
  - Southern Methodist University, Dallas, Texas
  - Baylor University, Waco, Texas

IPD SHARING:
Plan to Share IPD: Undecided